CLINICAL TRIAL: NCT02193477
Title: Effect of Transcutaneous Electrical Acupoint Stimulation (TEAS)on the Incidence Rate of Systemic Inflammatory Response Syndrome (SIRS) in Patients Undergoing Radical Surgery for Gastric Cancer
Brief Title: Effect of TEAS on the Incidence Rate of SIRS in Patients Undergoing Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, QiangWang,MD, associate professor,PhD advisor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Gjian
Record Dates: First submitted 2014-07-06; First posted 2014-07-17 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Systemic Inflammatory Response Syndrome; Inflammation
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Patients were given no TEAS.
- TEAS Treatment (Experimental): Patients were given 30min of TEAS before general anesthesia induction, 1th day and 2nd day after surgery.
  Interventions: Device: TEAS
- Sham TEAS (Sham Comparator): Patients were given 30min of sham TEAS before general anesthesia induction,1th day and 2nd day after surgery.
  Interventions: Device: Sham TEAS

INTERVENTIONS:
Device: TEAS — Electric stimulation was given through electrode attached to specific acupoints for 30mins before general anesthesia induction,1th day and 2nd day after surgery.
  Arms: TEAS Treatment
Device: Sham TEAS — Electric stimulation was given through electrode attached to non-acupoints for 30mins before general anesthesia induction,1th day and 2nd day after surgery.
  Arms: Sham TEAS

SUMMARY:
The purpose of this study is to access the effect of Transcutaneous Electrical Acupoint Stimulation(TEAS) on the Incidence rate of Systemic Inflammatory Response Syndrome (SIRS) in patients undergoing radical surgery for gastric cancer

DETAILED DESCRIPTION:
Patients undergoing elective radical surgery for gastric cancer under general anesthesia were randomly assigned to three groups, control group , TEAS group and sham TEAS group.

TEAS group receiving TEAS before general anesthesia induction , 1th day and 2nd day after surgery. TEAS was given through electrodes attached to specific acupoints. The time for TEAS was 30min.

Sham TEAS group receiving sham TEAS before general anesthesia induction , 1th day and 2nd day after surgery. Sham TEAS was given through electrodes attached to non-acupoints. The time for sham TEAS was also 30min.

Control group were given no TEAS. Incidence rates of SIRS in each group were compared .Venous blood samples from all groups(control group , TEAS group and sham TEAS group) were collected before general anesthesia induction,1th day and 3rd day after surgery. Inflammatory cytokines index including interleukin-6,interleukin-10,Tumor Necrosis Factor- alpha(TNF-α),Interferon-γ(IFN-γ),Monocyte Chemotactic Protein 1(MCP-1),IgG,IgM were measured.

ELIGIBILITY:
Inclusion Criteria:

* Age>30yrs,<75yrs
* ASA 1-2
* Scheduled for radical surgery for gastric cancer under general anesthesia；
* Informed consented

Exclusion Criteria:

* Patients with implanted pacemakers
* Patients with severe hypertension or cardiac dysfunction；
* Patients with severe pulmonary disease
* Patients with hemoglobin<90g/L

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of SIRS | 1st day after surgery
  SIRS is defined as 2 or more of the following variables :
  1. Fever of more than 38°C (100.4°F) or less than 36°C (96.8°F)
  2. Heart rate of more than 90 beats per minute
  3. Respiratory rate of more than 20 breaths per minute or arterial carbon dioxide tension (PaCO2) of less than 32mm Hg
  4. Abnormal white blood cell count (>12,000/µL or < 4,000/µL or >10% immature granulocyte forms)
  Incidence rate of SIRS is calculated using the following formula:
  (Number of SIRS Cases within the group) / (Number of Cases within the group)

SECONDARY OUTCOMES:
Change of Inflammatory cytokines | 30 minutes before general anesthesia induction and 1st and 3rd day after the surgery
  Venous blood samples were collected before general anesthesia induction,1th day and 3rd day after surgery. Inflammatory cytokines index including interleukin-6,interleukin-10,TNF-α,Interferon-γ(IFN-γ),Monocyte Chemotactic Protein 1(MCP-1),IgG,IgM were measured.
Incidence rate of SIRS | 3rd day after surgery
  SIRS is defined as 2 or more of the following variables :
  Fever of more than 38°C (100.4°F) or less than 36°C (96.8°F) Heart rate of more than 90 beats per minute Respiratory rate of more than 20 breaths per minute or arterial carbon dioxide tension (PaCO2) of less than 32mm Hg Abnormal white blood cell count (>12,000/µL or < 4,000/µL or >10% immature granulocyte forms)
  Incidence rate of SIRS is calculated using the following formula:
  (Number of SIRS Cases within the group) / (Number of Cases within the group)

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, MD, Study Chair — Air Force Military Medical University, China
Locations (1):
- Fourth Military Medical University, Xi’an, Shanxi, China